CLINICAL TRIAL: NCT07157553
Title: Effect of Argon Laser Panretinal Photocoagulation on Corneal Endothelial Cell Density Among Patients With Proliferative Diabetic Retinopathy .
Brief Title: Effect of Argon Laser Panretinal Photocoagulation on Corneal Endothelial Cell Density .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahlam Abdelhady Mohamad Omar, resident doctor at Ophthalmology department, Assiut University
Other Study IDs: argon laser photocoagulation
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Panretinal Photocoagulation
Keywords: panretinal photocoagulation; corneal endothelial cell density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population consists of 45 newly diagnosed patients of any age or sex with proliferative di: The inclusion criteria cover patients irrespective of age or sex who are newly diagnosed with proliferative diabetic retinopathy and are indicated for argon laser panretinal photocoagulation. Exclusion criteria include any history of corneal disease, previous intraocular surgeries, glaucoma, or intraocular inflammation to reduce confounding factors affecting corneal endothelial measurements. This helps to ensure that changes detected in corneal endothelial cell density and morphology are primarily attributable to the laser intervention rather than underlying ocular comorbidities. The sample size calculation determined that 45 patients would provide sufficient power to detect statistically significant changes, analyzed using paired t-tests and ANOVA for repeated measures.

SUMMARY:
This study investigates the effect of argon laser panretinal photocoagulation (PRP) on the corneal endothelial cell density (ECD) in patients with proliferative diabetic retinopathy (PDR) by comparing ECD measurements before and after PRP treatment.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is characterized by abnormal neovascularization driven by ischemic retinal tissue hypoxia and elevated vascular endothelial growth factor (VEGF) levels. Argon laser retinal photocoagulation (ALRP) is a standard treatment that applies thermal damage to the retinal pigment epithelium, reducing retinal oxygen demand and VEGF production, thereby causing regression of neovascular vessels. However, the laser light must pass through the anterior eye structures, potentially causing thermal and inflammatory damage to tissues such as the corneal endothelium, which is crucial for maintaining corneal transparency. This prospective observational clinical study conducted at Assuit University Hospital evaluates the impact of ALRP on corneal endothelial cell density using specular microscopy before, 1 week, and 1 month after PRP treatment in newly diagnosed PDR patients. Secondary outcomes include changes in cell morphology such as hexagonality and coefficient of variation, indicative of endothelial cell health and stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients from either sex with any age newly diagnosed PDR requring PRP .

Exclusion Criteria:

* history of corneal disease
* previous intraocular surgery
* glaucoma or intraocuar inflamation .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 45 newly diagnosed patients of any age or sex with proliferative diabetic retinopathy who require panretinal photocoagulation.
  The inclusion criteria cover patients irrespective of age or sex who are newly diagnosed with proliferative diabetic retinopathy and are indicated for argon laser panretinal photocoagulation. Exclusion criteria include any history of corneal disease, previous intraocular surgeries, glaucoma, or intraocular inflammation to reduce confounding factors affecting corneal endothelial measurements. This helps to ensure that changes detected in corneal endothelial cell density and morphology are primarily attributable to the laser intervention rather than underlying ocular comorbidities
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Endothelial Cell Density (ECD) after PRP | baseline
  The primary outcome is the quantitative change in the corneal endothelial cell density measured by specular microscopy, comparing pre-treatment baseline values with post-treatment values at 1 week and 1 month intervals. This measure reflects the potential impact of ALRP on the corneal endothelial integrity, crucial for corneal transparency and function.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212